CLINICAL TRIAL: NCT01254851
Title: Post Operative Walking Enhancements for Recovery (POWER) Trial
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Linda Brubaker, Professor, Dean, and Chief Diversity Officer, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 203031
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: External Causes of Morbidity and Mortality
Keywords: discharge criteria, gynecologic surgery, post-op ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- goal-augmented post-operative care. (Active Comparator): Patients in this group will be given a goal number of steps to take on each post-operative day.
  Interventions: Behavioral: goal-augmented post-operative care
- Usual care (No Intervention): routine post-operative ambulation

INTERVENTIONS:
Behavioral: goal-augmented post-operative care — Patients in the goal-augmented post-operative care group will be given a goal number of steps to take on each post-operative day following in-patient gynecologic surgery.
  Arms: goal-augmented post-operative care.

SUMMARY:
This study is a non-blinded randomized controlled trial. Consenting participants will be randomized to routine post-operative ambulation vs. goal-augmented post-operative care (they will be given a goal number of steps to take on each post-operative day) following in-patient gynecologic surgery.

DETAILED DESCRIPTION:
This study is a non-blinded randomized controlled trial. Consenting participants will be randomized to routine post-operative ambulation vs. treadmill-augmented post-operative care (placement of non-motorized treadmill in their room) following in-patient gynecologic surgery.

We will approach all women undergoing gynecologic procedures that are expected to ambulate within 12 hours of their operation and are anticipated to remain hospitalized at least 18 hours. Following confirmation of eligibility, we will enroll subjects either in the clinic when they are being consented for their gynecologic procedure or upon presentation to the hospital the day of their procedure. Randomization will occur at the completion of the gynecologic procedure when it has been confirmed by the primary surgeon that the patient is able to ambulate independently within 12 hours after completion of the procedure. At that time, participants will be randomized using opaque envelopes prepared by the study statistician in a 1:1 ratio to receive usual post-operative care or treadmill-augmented care.

All patients will have a pedometer placed on their person in the post-anesthesia recovery unit (PACU) which will be removed the day of their discharge. The primary outcome assessed will be number of steps taken in the 24 hour period prior to discharge as assessed by the electronic pedometer readings.

Pedometer will be placed on patients using a lanyard and pedometer clip in the recovery room. No participant will start ambulation without physician's clinical order. When the patient is ready for the first ambulation she will be accompanied by a nurse to sit up in a chair. Once the patient is able to ambulate herself she may ambulate in her room or in the hallway or if randomized to treadmill group she will be able to ambulate on the treadmill. She will be wearing her pedometer at all times until discharge from Loyola.

ELIGIBILITY:
Inclusion Criteria:

* Independent ambulation pre-operatively
* Undergoing gynecologic procedure
* Expected to ambulate within 12 hours of their procedure

Exclusion Criteria:

* Children under the age of 18
* Inability to ambulate independently prior to their surgery
* Primary surgeon does not want patient to ambulate within 12 hours of procedure
* English is not the primary language spoken by the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Brubaker, M.D., Principal Investigator — Loyola University
Locations (2):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - Gottlieb Memorial Hospital, Melrose Park, Illinois

REFERENCES:
- [Derived] Liebermann M, Awad M, Dejong M, Rivard C, Sinacore J, Brubaker L. Ambulation of hospitalized gynecologic surgical patients: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):533-537. doi: 10.1097/AOG.0b013e318280d50a. PMID 23635615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized controlled trial enrolled patients who were going to undergo gynecologic surgery were enrolled from 1/11-6/11 at Loyola University Medical Center .We approached adult (>18 years) English speaking women prior to undergoing major gynecologic surgery who were expected to have at least a 24-hour hospital stay post-operatively.
Pre-assignment Details: All Enrolled patients were randomized to a group. Those patients who were enrolled but not included in statistical analysis had their data lost due to lost pedometer.
Period: Overall Study
Arm/Group | Goal-augmented Post-operative Care. | Usual Care
Started | 69 | 77
Completed | 61 | 68
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal-augmented Post-operative Care. | Usual Care | Total
Number analyzed (Participants) | 69 | 77 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 61 | 114
  >=65 years | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.1) | 53.9 (13.27) | 54.98 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 77 | 146
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 77 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Steps Taken in 24 Hours.
Description: The primary outcome assessed was the number of steps taken in the 24 hour period prior to discharge as assessed by the electronic pedometer readings.
Time Frame: 1 day
Population: The analysis is an intention to treat (ITT) analysis comprising all participants who were randomized.
Measure: Median (Full Range); unit: Steps
Arm/Group | Goal-augmented Post-operative Care. | Usual Care
Number analyzed (Participants) | 69 | 77
Steps | 80 [0 to 2353] | 87 [0 to 3576]
Statistical Analysis 1: Comparison: Goal-augmented Post-operative Care. vs Usual Care; Test type: Superiority or Other; p = .70, Wilcoxon (Mann-Whitney); Standardized test statistic (z-score) = 0.39

ADVERSE EVENTS:
Time Frame: During Hospitalization.
Arm/Group | Goal-augmented Post-operative Care. | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/77
Other Adverse Events (participants affected / at risk) | 0/69 | 0/77

LIMITATIONS AND CAVEATS:
Difficulty ensuring that encouragement was given, as we did not quantify the frequency of encouragement by the health care team. Loss of data due to loss of pedometers

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes